CLINICAL TRIAL: NCT02393378
Title: A 24-week Randomized, Open-Label, Parallel-Group, Active-Controlled, Exploratory, Proof-of-Mechanism Imaging Study Investigating the Efficacy of 150 mg of Namilumab Administered Subcutaneously vs Adalimumab in Patients With Moderate to Severe Early Rheumatoid Arthritis Inadequately Responding to Methotrexate
Brief Title: Namilumab vs Adalimumab in Participants With Moderate to Severe Early Rheumatoid Arthritis Inadequately Responding to Methotrexate
Acronym: TELLUS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision - to understand data from psoriasis study - NCT02129777 and wait for results of formal proof of concept study - NCT02379091.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT203-2004; U1111-1160-1791 (Registry Identifier: WHO); 15/SC/0020 (Registry Identifier: NRES); 2014-002945-23 (EudraCT Number); REec-2015-1508 (Registry Identifier: REec)
Record Dates: First submitted 2015-03-15; First posted 2015-03-19 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2018-08

CONDITIONS: Rheumatoid Arthritis
Keywords: Drug Therapy
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — namilumab; Adalimumab; Methotrexate; Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adalimumab 40 mg (Experimental): Adalimumab 40 mg, subcutaneous (SC) injection at Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 22 as an add-on to weekly existing stable MTX and folic acid as per prescribed medication.
  Interventions: Drug: Adalimumab; Drug: Methotrexate; Drug: Folic Acid
- Namilumab 150 mg (Active Comparator): Namilumab 150*2 mg, SC injection at Week 0 followed by 150 mg, SC injections at Weeks 2, 6, 10, 14, 18, and 22 as an add-on to weekly existing stable MTX and folic acid as per prescribed medication.
  Interventions: Drug: Namilumab; Drug: Methotrexate; Drug: Folic Acid

INTERVENTIONS:
Drug: Namilumab — Namilumab injection
  Arms: Namilumab 150 mg
Drug: Adalimumab — Adalimumab SC injection
  Arms: Adalimumab 40 mg
Drug: Methotrexate — Methotrexate tablet
Drug: Folic Acid — Folic Acid Tablet

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of namilumab in combination with existing methotrexate (MTX) therapy over 24 weeks in participants with moderate to severe early rheumatoid arthritis (RA), diagnosed within 6 months and inadequately controlled by MTX alone.

DETAILED DESCRIPTION:
The drug being investigated in this study is namilumab for the treatment of moderate to severe Rheumatoid Arthritis (RA). This study will evaluate the efficacy and safety of namilumab in participants diagnosed with RA within 6 months and insufficiently controlled by methotrexate (MTX) alone.

The study will enroll approximately 36 patients, who will be randomly assigned in a 2:1 ratio to the following open label treatment groups:

* Namilumab 150 mg + MTX + folic acid
* Adalimumab 40 mg + MTX + folic acid

Imaging techniques, including Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI), will be used to measure changes in the dominant hand and the wrist.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is a maximum of 42 weeks, including follow-up period. Participants will make 16 visits to the site and will be followed up by telephone twice after end of treatment.

A strategic decision was made to stop the study on 18 December 2015 in order to fully understand the data from the psoriasis study (ClinicalTrials.gov Identifier:NCT02129777) and wait for the results of the formal proof of concept study (ClinicalTrials.gov Identifier: (NCT02379091) in participants with rheumatoid arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Is diagnosed with adult onset rheumatoid arthritis (RA) as defined by the 2010 The American College of Rheumatology (ACR)/The European League Against Rheumatism criteria for the classification of RA within 6 months prior to Screening Visit.
* Has active disease defined as:

  1. swollen joint count ≥4 and tender joint count ≥4 (referred to the 28 joint-count system) at Screening and Baseline Visits, and
  2. C-reactive protein ≥4.3 mg/L and erythrocyte sedimentation rate ≥28 mm/hr at Baseline Visits, and
  3. imaging (ultrasound power doppler) evidence of moderate to severe inflammation of at least 1 joint of the dominant hand metacarpophalangeal (MCP) and/or wrist) at Screening and Baseline Visits.
* Is receiving current treatment with Methotrexate (MTX) for RA.
* Received MTX for at least 3 months prior to the Screening Visit.
* Received treatment with MTX ≥15 to 25 mg/week at a stable dose via the same route of administration and formulation for at least 8 weeks prior to the Baseline Visit, OR
* Participants on a stable dose for at least 8 weeks of MTX of ≥7.5 mg/week, if the MTX dose has been reduced for reasons of documented intolerance to MTX.
* Is willing to continue or initiate treatment with oral folic acid (at least 5 mg/week) or equivalent and be treated during the entire trial (mandatory co-medication for MTX treatment).
* Has a posterior, anterior, and lateral chest x-ray obtained within the last 3 months before Screening or at the Screening visit without any signs of clinically significant pulmonary disease.

Exclusion Criteria:

* Has received biologic disease-modifying antirheumatic drugs for the treatment of RA.
* Have a history of or currently inflammatory joint disease other than RA (e.g., gout, reactive arthritis, psoriatic arthritis, seronegative spondyloarthropathy, or Lyme disease) or other systemic autoimmune disorder (eg, systemic lupus erythematosus, inflammatory bowel disease, scleroderma, inflammatory myopathy, mixed connective tissue disease, or other overlap syndrome).
* Has any major systemic features of RA, for example, Felty's syndrome, vasculitis, or interstitial fibrosis of the lungs.
* Diagnosed with primary fibromyalgia that would make it difficult to appropriately assess RA activity for the purposes of this study or a diagnosis of any systemic inflammatory condition other than RA.
* Has a history of juvenile idiopathic arthritis or RA onset prior to age 16 years.
* Required to take excluded medications
* Not willing to take folic/folinic acid (as part of MTX regimen, according to country-specific practices) in order to minimize toxicity.
* Has an underlying condition that predisposes to infections (e.g., immunodeficiency, poorly controlled diabetes history, splenectomy).
* Has a history of clinically significant interstitial lung disease, for example, history of chronic or recurrent pulmonary infection where macrophages are important for the clearance of the infection, for example, pneumocystis carinii pneumonia, allergic bronchopulmonary aspergillosis, nocardia infections, Actinomyces infection.
* Presence or history of active tuberculosis (TB) or latent TB infection, where no anti-TB treatment has been given or where successful completion of an appropriate course of anti-TB therapy cannot be documented.
* A positive QuantiFERON-TB Gold test and/or evidence of active or latent TB by chest x-ray at Screening Visit, not accompanied by initiation of an approved regimen of anti-TB therapy at least 12 months prior to the Baseline Visit.
* Has a known history of infection with hepatitis B virus, hepatitis C virus, or human immunodeficiency virus (HIV), or has serological findings at the Screening Visit which indicate active or latent hepatitis B, hepatitis C or HIV infection.
* Has a clinically relevant decrease in lung function at Screening, as defined by an oxygen saturation as measured by pulse oximetry (SpO2) <94% at rest.
* Has evidence of clinically significant respiratory disease on the basis of review the data from participants' respiratory assessments including chest x-ray, pulmonary function test (forced expiratory volume in 1 second [FEV1] and forced vital capacity [FVC]) by spirometry performed at Screening). The participants must have SpO2 ≥94%, FEV1 and/or FVC ≥60% of predicted values at Screening or at Baseline and no uncontrolled lung disease. Participant's treatment that has been modified to control lung disease within 24 weeks prior to Screening is exclusionary.
* Has a history of severe chronic obstructive pulmonary disease (COPD) and/or history of severe COPD exacerbation(s), or a history of asthma with exacerbations requiring hospitalization, within the last 12 months prior to the Screening Visit.
* Has an estimated glomerular filtration rate (eGFR) of less than 60 mL/min/1.73m2.History of MTX-associated lung toxicity.
* Has a history or evidence of a clinically significant disorder (including but not limited to cardiopulmonary, oncologic, renal, metabolic, hematologic or psychiatric), condition or disease that, in the opinion of the investigator and Takeda physician, would pose a risk to participant safety or interfere with the study evaluation, procedures or completion.
* Has any significant cardiac disease (eg, coronary artery disease with unstable angina, coronary heart failure New York Heart Association Class III and IV, familial long QT syndrome).
* Has a history of cancer within the last 10 years except for basal cell or squamous cell carcinomas of the skin or in situ carcinoma of the cervix treated and considered cured.
* Has a severe psychiatric or neurological disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (13):
- Czechia (2):
  - Pardubice
  - Prague
- Estonia (2):
  - Tallinn
  - Tartu
- Russia (2):
  - Moscow
  - Yaroslavl
- Spain (4):
  - Santiago de Compostela, La Coruna
  - Fuenlabrada, Madrid
  - A Coruña
  - Madrid
- United Kingdom (3):
  - London, Greater London
  - Salford, Greater Manchester
  - Oxford, Oxfordshire

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 5 investigative sites in Estonia and Russian Federation from 08 April 2015 to 03 November 2016.
Pre-assignment Details: Participants with a diagnosis of rheumatoid arthritis were enrolled in 2:1 ratio to receive either namilumab combined with methotrexate (MTX) or adalimumab combined with MTX.
Groups:
- Adalimumab 40 mg: Adalimumab 40 mg SC injection at Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, and 22 as an add-on to weekly existing stable MTX and folic acid as prescribed in clinical practice.
- Namilumab 150 mg: Namilumab 300 mg SC injection at Week 0 followed by 150 mg SC injection at Weeks 2, 6, 10, 14, 18, and 22 as an add-on to weekly existing stable MTX and folic acid as prescribed in clinical practice.
Period: Overall Study
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (7.21) | 61.3 (6.90) | 62.0 (6.48)
Age, Customized [Count of Participants; unit: Participants]
  45 to 64 years | 1 | 3 | 4
  >= 65 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 4 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  Estonia | 1 | 2 | 3
  Russia | 2 | 2 | 4
Height [Mean (Standard Deviation); unit: cm] | 171.7 (8.96) [88.0 to 117.0] | 162.5 (3.00) [60.0 to 99.2] | 166.4 (7.44) [60.0 to 117.0]
Weight [Mean (Standard Deviation); unit: kg] | 106.67 (16.197) [26.6 to 42.0] | 78.83 (16.550) [22.3 to 36.2] | 90.76 (21.116) [22.3 to 42.0]
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = Weight in kg/Height in square meters.
  kg/m^2 | 36.77 (8.806) | 29.68 (5.844) | 32.71 (7.569)
Body Mass Index (BMI) Categories [Count of Participants; unit: Participants]
  < 30 kg/m^2 | 1 | 2 | 3
  >= 30 kg/m^2 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Synovitis, Erosion and Bone Marrow Edema (Osteitis) Score at Week 24
Description: A Magnetic Resonance Imaging (MRI) of Metacarpophalangeal (MCP) and Wrist of the dominant hand was performed at the baseline and at week 24. Change from the Baseline was assessed according to the Outcome Measures in Rheumatoid Arthritis (RA) Clinical Trials RA-MRI scoring (OMERACT RAMRIS) Standard. RAMRIS score is the sum of its core components: Synovitis Score, Edema Score, and Erosion Score. Synovitis is scored from 0 (normal) to 9 (maximum distension of synovial cavity). Edema is scored 0 (normal) to 69 (maximum articular bone involvement). Erosion is scored from 0 (normal) to 230 (maximum erosion of articular bone). Total RAMRIS score=0 (normal), maximum RAMRIS score=308 (severe structural damage). For Synovial Score, Edema Score, Erosion Score, and RAMRIS score, increasing number = increasing severity.
Time Frame: Baseline and Week 24
Population: Full analysis set included participants who received at least one dose of study medication. Here number analyzed is the number of participants who were evaluated for specific sub-score.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Number analyzed (Participants) | 3 | 4
score on a scale
  Erosion Score, Change at Week 24: number analyzed (Participants) | 3 | 3
  Erosion Score, Change at Week 24 | 0.50 (0.866) | 0.00 (0.500)
  Synovitis Score, Change at Week 24: number analyzed (Participants) | 3 | 3
  Synovitis Score, Change at Week 24 | 0.17 (0.764) | -1.50 (4.770)
  Osteitis Score, Change at Week 24: number analyzed (Participants) | 3 | 2
  Osteitis Score, Change at Week 24 | -0.33 (0.764) | -2.00 (3.536)

2. Secondary Outcome: Change From Baseline in Dynamic Contrast-enhanced - Magnetic Resonance Imaging (DCE-MRI) Parameters at Week 24
Description: DCE-MRI was used to measure synovial vascular perfusion. The change from baseline in DCE-MRI parameters of synovial vascular perfusion at Week 24 were measured.
Time Frame: Baseline and Week 24
Population: Full analysis set included participants who received at least one dose of study medication. Hence, number analyzed is the number of participants who were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Number analyzed (Participants) | 3 | 3
mL | 0.016 (0.0253) | -0.052 (0.0662)

3. Secondary Outcome: Number of Participants Who Achieved Remission at Week 24
Description: Remission is defined as the number of participants who achieved Disease Activity Score 28 based on C-reactive protein (DAS28-CRP) score <2.6. The DAS28-CRP is a composite measure of inflammation in rheumatoid arthritis (RA) and incorporates a tender and swollen joint count, CRP and patient global assessment of disease activity expressed in a gaussian distribution of variables ranging from 0 to 10. A DAS28-CRP score of <3.2 suggests a low level of disease activity, while a score of >5.1 suggests a high level of disease activity. Using the DAS-CRP as a continuous scale allows investigators (and clinicians) to measure a clinically meaningful endpoint following institution of a therapeutic intervention. In RA, clinical remission would therefore be graded as a DAS28 score of ≤2.6 with disease flare accompanying scores of ≥5.1; well-controlled disease is best characterized as fitting in between these two scores.
Time Frame: Week 24
Population: Full analysis set included participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Number analyzed (Participants) | 3 | 4
Participants | 0 | 2

4. Secondary Outcome: Number of Participants Who Achieved Low Disease Activity at Week 24
Description: Disease Activity Score 28 based on C-reactive protein (DAS28-CRP) low disease activity is defined as a score <3.2. The DAS28-CRP is a composite measure of inflammation in RA and incorporates a tender and swollen joint count, CRP and patient global assessment of disease activity expressed in a gaussian distribution of variables ranging from 0 to 10. A DAS28-CRP score of <3.2 suggests a low level of disease activity, while a score of >5.1 suggests a high level of disease activity. Using the DAS-CRP as a continuous scale allows investigators (and clinicians) to measure a clinically meaningful endpoint following institution of a therapeutic intervention. In RA, clinical remission would therefore be graded as a DAS28 score of ≤2.6 with disease flare accompanying scores of ≥5.1; well-controlled disease is best characterized as fitting in between these two scores.
Time Frame: Week 24
Population: Full analysis set included participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Number analyzed (Participants) | 3 | 4
Participants | 2 | 4

5. Secondary Outcome: Number of Participants Who Achieved ACR 20, 50, and 70 at Week 24
Description: The American College of Rheumatology (ACR) 20 is composite index of improvement in RA proposed by the ACR. ACR20 refers to a composite improvement of 20% in swollen joint count, tender joint count, and 3 or more of the following 5 measures: Physician's Global Assessment of Disease Activity, Patient's Global Assessment of Disease Activity, Patient Pain VAS, Patient's self-addressed disability (HAQ), Acute-phase reactant (ESR or CRP) The ACR 50 and ACR 70 are similar tools, used to indicate 50% and 70% improvement, respectively.
Time Frame: Week 24
Population: Full analysis set included participants who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Number analyzed (Participants) | 3 | 4
Participants
  ACR 20 | 2 | 4
  ACR 50 | 2 | 3
  ACR 70 | 1 | 2

6. Secondary Outcome: Change From Baseline in DAS28-CRP Score
Description: The DAS28-CRP is a composite measure of inflammation in RA and incorporates a tender and swollen joint count, CRP and patient global assessment of disease activity expressed in a gaussian distribution of variables ranging from 0 to 10. A DAS28-CRP score of <3.2 suggests a low level of disease activity, while a score of >5.1 suggests a high level of disease activity. Using the DAS-CRP as a continuous scale allows investigators (and clinicians) to measure a clinically meaningful endpoint following institution of a therapeutic intervention. In RA, clinical remission would therefore be graded as a DAS28 score of ≤3.2 with disease flare accompanying scores of ≥5.1; well-controlled disease is best characterized as fitting in between these two scores.
Time Frame: Baseline Up to Week 42
Population: Full analysis set included participants who received at least one dose of study medication. Here number analyzed is the number of participants who were evaluated at specific time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Number analyzed (Participants) | 3 | 4
score on a scale
  Week 2: number analyzed (Participants) | 2 | 3
  Week 2 | -0.55 (0.737) | -0.78 (0.333)
  Week 6 | -1.36 (1.086) | -1.58 (0.494)
  Week 10: number analyzed (Participants) | 2 | 4
  Week 10 | -1.74 (1.103) | -1.83 (0.344)
  Week 12 | -1.94 (1.036) | -2.12 (0.613)
  Week 18 | -2.05 (1.136) | -2.72 (0.486)
  Week 24 | -2.04 (1.596) | -2.99 (0.216)
  Week 32 | -1.89 (1.946) | -2.38 (0.862)
  Week 42 | -1.99 (1.938) | -1.57 (1.387)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 42
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Adalimumab 40 mg | Namilumab 150 mg
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg (N=3) | Namilumab 150 mg (N=4)
Cellulitis streptococcal (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg (N=3) | Namilumab 150 mg (N=4)
Streptococcal sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Forced expiratory volume decreased (Investigations) | 0 | 1
Forced vital capacity decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.